CLINICAL TRIAL: NCT00243906
Title: Interventional Management of Stroke (IMS) II Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01NS039160 (NIH)
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Stroke
Keywords: acute ischemic stroke; stroke; rt-PA; thrombolytic; recombinant tissue plasminogen activator
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Tissue Plasminogen Activator; Ultrasonic Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Recombinant tissue plasminogen activator — Low-dose IV rt-PA (0.6 mg/kg) followed by delivery of additional IA rt-PA (up to 22 mg).
Procedure: Low-intensity ultrasound — Delivery of additional IA rt-PA (up to 22 mg) in the setting of low-energy ultrasound via the EKOS microinfusion catheter at the site of IA occlusion in acute ischemic stroke patients with large strokes (NIHSS >/= 10) treated within 3 hours of symptoms onset.

SUMMARY:
The purpose of this study is to examine the effects of delivering intra-arterial recombinant tissue plasminogen activator (rt-PA) and ultrasound to the site of the blood clot blocking blood flow to the brain of stroke patients.

DETAILED DESCRIPTION:
The overall goal of Interventional Management of Stroke (IMS II) study is to refine thrombolytic therapy for patients with acute ischemic stroke who can be treated within three hours of stroke onset.

This multi-center, non-randomized pilot study will provide preliminary data about the benefits and risks of combined intravenous (IV) and intra-arterial (IA) recombinant tissue plasminogen activator (rtPA) and low-intensity ultrasound energy in ischemic stroke patients with baseline NIHSSS >/= 10 in whom intravenous treatment can be started within three hours of stroke onset. rt-PA is a thrombolytic, clot-dissolving drug.

The primary objectives for the study are to obtain reliable estimates of the effectiveness and safety of a treatment approach combining IV/IA rt-PA and ultrasound for stroke patients; and to determine if the estimated effectiveness of combined IV/IA rt-PA at 3 months-as compared to the 3 month outcome of placebo-treated patients in the NINDS rt-PA Stroke Trial-warrants proceeding to a large, phase III randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 through 80 years (i.e., candidates must have had their 18th birthday, but not had their 81st birthday)
* Initiation of intravenous rt-PA within 3 hours of onset of stroke symptoms. Time of onset is defined as the last time when the subject was witnessed to be at baseline (i.e., subjects who have stroke symptoms upon awakening will be considered to have their onset at beginning of sleep)
* An NIHSSS >/= 10 at the time that intravenous rt-PA is begun

Exclusion Criteria:

* History of stroke in the past 3 months
* Previous intra-cranial hemorrhage, neoplasm, subarachnoid hemorrhage, or arteriovenous malformation
* Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT scan is normal
* Hypertension at time of treatment; systolic BP > 185 or diastolic > 110 mm Hg) or aggressive measures to lower blood pressure to below these limits are needed.
* Presumed septic embolus
* Presumed pericarditis, including pericarditis after acute myocardial infarction
* Recent (within 30 days) surgery or biopsy of parenchymal organ
* Recent (within 30 days) trauma, with internal injuries or ulcerative wounds
* Recent (within 90 days) severe head trauma or head trauma with loss of consciousness
* Any active or recent (within 30 days) hemorrhage
* Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency or oral anticoagulant therapy with INR > 1.5 or institutionally equivalent prothrombin time
* Females of childbearing potential who are known to be pregnant and/or lactating or who have positive pregnancy tests on admission
* Baseline lab values: glucose < 50mg/dl or > 400mg/dl, platelets <100,000, or Hct <25
* Subjects that require hemodialysis or peritoneal dialysis
* Subjects who have received heparin within 48 hours must have a normal partial thromboplastin time (PTT) to be eligible
* Subjects with an arterial puncture at a non-compressible site or a lumbar puncture in the previous 7 days
* Subjects with a seizure at onset of stroke
* Subjects with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations
* Other serious, advanced, or terminal illness
* Any other condition that the investigator feels would pose a significant hazard to the subject if Activase (Alteplase) therapy is initiated
* Current participation in another research drug treatment protocol; subject cannot start another experimental agent until after 90 days
* Informed consent is not or cannot be obtained. For example, obtunded subjects are not automatically excluded from the study. However, if the next of kin or legal guardian (i.e., the individual legally empowered in the state where the consent is obtained) cannot provide consent, randomization and entry into the study could not proceed

CT Scan Exclusion Criteria:

* High density lesion consistent with hemorrhage of any degree
* Significant mass effect with midline shift
* Large (more than 1/3 of the middle cerebral artery) regions of clear hypodensity on the baseline CT scan. Sulcal effacement and/or loss of grey-white differentiation alone are not contraindications for treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2003-01; Primary Completion 2006-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 36 hours after completion of rt-PA infusion
  Development of intracerebral hematoma or hemorrhagic infarction with clinical deterioration likely to result in permanent disability or death, or other severe systemic bleeding complications such as groin hematoma, retroperitoneal hematoma, or gastrointestinal bleeding requiring transfusion of 3 units of blood replacement or major surgical intervention.
Primary Angiographic Outcome | 60 minutes after start of IA therapy
  The primary revascularization end point was complete (arterial occlusive lesion III) recanalization of the targeted arterial occlusion at 60 minutes after the start of IA rt-PA and ultrasound therapy,
Primary Outcome Measure | 3 months following treatment
  modified Rankin Score of 0 or 1

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P. Broderick, MD, Principal Investigator — University of Cincinnati; Thomas A. Tomsick, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Background] IMS II Trial Investigators. The Interventional Management of Stroke (IMS) II Study. Stroke. 2007 Jul;38(7):2127-35. doi: 10.1161/STROKEAHA.107.483131. Epub 2007 May 24. PMID 17525387